CLINICAL TRIAL: NCT02941445
Title: Weight Maintenance With Dipeptidyl Peptidase 4 (DPP4) Inhibitor Sitagliptin in Combination With Metformin After Liragludite Induced Weight Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Andrej Janez, MD PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SITA after LIRA
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Polycystic Ovary Syndrome; Body Weight
Keywords: DPP4-inhibitors
MeSH Terms: conditions — Polycystic Ovary Syndrome; Body Weight | interventions — Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- COMBO (sitagliptin and metformin) (Experimental): metformin 1000 mg BID and sitagliptin 50mg BID for 12 weeks
  Interventions: Drug: sitagliptin and metformin
- MET (metformin) (Experimental): metformin 1000 mg BID
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: sitagliptin and metformin
  Other Names: Janumet
  Arms: COMBO (sitagliptin and metformin)
Drug: Metformin
  Other Names: Glucophage
  Arms: MET (metformin)

SUMMARY:
Weight reduction is the most important treatment target in obese women with polycystic ovary syndrome (PCOS), yet it is usually hardly achievable with lifestyle intervention alone. Glucagon-like peptide 1 (GLP-1) receptor agonist (RA) liraglutide was recently approved as an anti-obesity drug but with some limitations, which include high cost and the lack of long-term efficacy and safety data regarding weight reduction. In addition, weight loss achieved with liraglutide is often non-sustainable after treatment cessation. Although DPP-4 inhibitors are weight neutral, they reduced weight regain in animals previously treated with GLP-1 RAs if they were switched to DPP-4 inhibitor rather than placebo. The aim is to evaluate whether DPP-4 inhibitor sitagliptin in combination with metformin reduce body weight regain more effectively than metformin alone in obese PCOS who had been previously treated with liraglutide.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old to menopause
* polycystic ovary syndrome (NICHD criteria)
* BMI of 30kg/m2 or higher

Exclusion Criteria:

* type 1 or type 2 diabetes mellitus
* history of carcinoma
* Cushing's syndrome or congenital (non-classic) adrenal hyperplasia
* personal or family history of multiple endocrine neoplasia type 2
* significant cardiovascular, kidney or hepatic disease
* the use of statins, within 90 days prior to study entry

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in body weight. | Patient's body weight was measured at the baseline and after 12 weeks of clinical trial.

SECONDARY OUTCOMES:
Change in body mass indey (BMI). | Patient's body height was measured at the baseline. Body weight was measured at the baseline and after 12 weeks of clinical trial.
  The BMI was calculated as the body mass divided by the square of the body height (kg/m2)

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janež, MD PhD, Principal Investigator — University Medical Centre Ljubljana

IPD SHARING:
Plan to Share IPD: No